CLINICAL TRIAL: NCT03752463
Title: NMDA Enhancer for the Treatment of Mild Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 105-3412C
Record Dates: First submitted 2018-11-21; First posted 2018-11-26 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- DAOI-A group (Experimental)
  Interventions: Drug: DAOI-A group
- DAOI-B group (Experimental)
  Interventions: Drug: DAOI-B group
- DAOI-C group (Experimental)
  Interventions: Drug: DAOI-C group
- Placebo group (Placebo Comparator)
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: DAOI-A group — DAOI with A dose
  Arms: DAOI-A group
Drug: DAOI-B group — DAOI with B dose
  Arms: DAOI-B group
Drug: DAOI-C group — DAOI with C dose
  Arms: DAOI-C group
Drug: Placebo oral capsule — Placebo
  Arms: Placebo group

SUMMARY:
NMDA neurotransmission plays an important role in learning and memory. NMDA receptors (NMDAR) were found to decrease in the frontal lobe and hippocampus of Alzheimer's disease (AD). This study is a randomized, double-blind, placebo controlled drug trial for testing the efficacy of NMDAR-enhancer. All subjects will be allocated randomly to 4 groups: (1) DAOI-A group; (2) DAOI-B group; (3) DAOI-C group; (4) placebo group. The study period is 24 weeks. The investigators hypothesize that DAOI may yield better efficacy than placebo for cognitive function in patients with AD.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Alzheimer's disease
* MMSE between 10-26
* CDR 1

Exclusion Criteria:

* Hachinski Ischemic Score > 4
* Substance abuse/dependence
* Parkinson disease, epilepsy, dementia with psychotic features
* Major depressive disorder
* Major physical illnesses
* Severe visual or hearing impairment

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2015-05-22 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the Alzheimer's disease assessment scale - cognitive subscale at week 8, 16 and 24 | week 0, 8, 16, 24
  Cognitive assessment

SECONDARY OUTCOMES:
Change from baseline in Clinician's Interview-Based Impression of Change plus Caregiver Input at week 8, 16 and 24 | week 8, 16, 24
  Global assessment
Change from baseline in speed of processing (Category Fluency) at week 24 | week 0, 24
  Cognitive assessment
Change from baseline in working memory (Wechsler Memory Scale, Spatial Span) at week 24 | week 0, 24
  Cognitive assessment
Change from baseline in verbal learning and memory tests (Wechsler Memory Scale, Word Listing) at week 24 | week 0, 24
  Cognitive assessment

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

REFERENCES:
- [Derived] Lin CH, Lane HY. Sodium benzoate treatment decreased amyloid beta peptides and improved cognitive function among patients with Alzheimer's disease: secondary analysis of a randomized clinical trial. Transl Psychiatry. 2025 Aug 5;15(1):264. doi: 10.1038/s41398-025-03492-3. PMID 40764372
- [Derived] Lane HY, Wang SH, Lin CH. Sex- and dose-dependent catalase increase and its clinical impact in a benzoate dose-finding, randomized, double-blind, placebo-controlled trial for Alzheimer's disease. Pharmacol Biochem Behav. 2024 Dec;245:173885. doi: 10.1016/j.pbb.2024.173885. Epub 2024 Oct 9. PMID 39384087